CLINICAL TRIAL: NCT02769728
Title: EndoBarrierTM in Obese Subjects With Type 2 Diabetes: Impact on Pancreatic Function, Insulin Resistance, Gut Peptides and Gut Permeability - a Pilot Study
Brief Title: EndoBarrier in Obese Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2014-01
Record Dates: First submitted 2016-05-03; First posted 2016-05-12 (Estimated); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: The endobarrier device was implanted and explanted under general anaesthesia by trained gastroenterologists.
Masking Description: no masking
Oversight: Data Monitoring Committee: No

ARMS (1):
- EndoBarrier (Experimental): EndoBarrier will be implemented for 9 months.
  Interventions: Device: EndoBarrier

INTERVENTIONS:
Device: EndoBarrier — implantation of a duodeno-jejunal bypass liner for weight reduction in obese subjects with type 2 diabetes mellitus
  Other Names: duodeno-jejunal bypass liner

SUMMARY:
The aim of the study is to explore short and longer-term effects of the Endobarrier™ implantation on insulin resistance and beta-cell function assessed by repeated Botnia clamps. In addition changes in gut peptides and gut permeability after implantation of a removable duodeno-jejunal bypass device to induce diabetes remission in obese subjects with sub-optimally controlled type 2 diabetes mellitus will be determined. Further changes in body weight and body composition, the change in global cardiovascular risk from baseline to 12 months, estimated using the UKPDS risk engine will be recorded.

DETAILED DESCRIPTION:
Obesity and diabetes probably represent the most challenging threat to public health in the 21st century. Obesity has multiple deleterious effects on health, significantly increasing the risk of fatal and non-fatal diseases including type 2 diabetes (T2DM). Bariatric surgery is a well-established method for the treatment of morbid obesity and has increasingly been recognized as an effective, long-lasting treatment option for T2DM.

Recently a potential, non-invasive alternative to bariatric surgery, a duodenal-jejunal bypass liner (EndoBarrierTM) has been introduced. It is an endoscopically implantable and removable device that prevents contact between partially digested nutrients and the proximal intestine. This device was shown to reduce body weight and to improve glycaemic control in subjects with diabetes. Small pilot studies suggested a change in incretin levels, similar to that observed after gastric surgery with an improvement of insulin sensitivity and glucose metabolism. To better understand and characterize the hormonal and/or metabolic effects after the implantation and removal of the EndoBarrierTM, this monocentric, prospective, trial is being performed.

The primary objective of this study is to clarify the changes in gut peptides and gut permeability after implantation the EndoBarrierTM in obese subjects with sub-optimally controlled type 2 diabetes mellitus. Additionally, the investigators aim to determine the changes in body weight and measure of adiposity, the change in global cardiovascular risk from baseline to 12 months as well as the changes in insulin sensitivity and beta-cell function over time.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Type 2 diabetes
* BMI 30-49 kg/m²
* HbA1c ≥ 6.5% (48 mmol/mol)
* Appropriate life style intervention measures have been tried but have failed to achieve or maintain adequate, clinically beneficial weight loss for at least 6 months
* Person is generally fit for intervention
* Person commits to the need for long-term follow-up

Exclusion Criteria:

* Type 1 diabetes mellitus
* Maturity Onset Diabetes of the Young (MODY)
* Secondary diabetes due to a specific disease or glucocorticoid therapy
* Pregnancy or women of childbearing age without adequate contraception
* Women who are breast-feeding
* Hypothalamic cause of obesity, Cushing syndrome
* Major psychiatric disease including diagnosed eating disorders, history of drug or alcohol abuse
* History of bariatric surgery or complex abdominal surgery
* Inflammatory bowel disease
* Pancreatitis
* Cholelithiasis
* Uncontrolled gastroesophageal reflux
* Known upper GI bleeding conditions, e.g. gastric or esophageal varices
* Congenital or acquired abnormalities of the upper GI tract, e.g. stenosis
* Subjects with or a history of coagulopathy, upper gastro-intestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasia
* Chronic non-steroidal anti-inflammatory drug (NSAID) or aspirin treatment (Subjects unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during the implant period)
* Previous GI surgery that could affect the ability to place the device or the function of the implant
* GLP-1 receptor agonist therapy
* Known ischaemic heart disease or heart failure
* History of stroke
* Active Helicobacter pylori (Note: Subjects may be enrolled if they had a prior history of Helicobacter Pylori and were successfully treated)
* Iron deficiency and/or iron deficiency anemia
* Subjects or Family history of a known diagnosis or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
* Known malignancy or any other multimorbid patient condition or circumstance, which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol or would put the participant at an unjustified risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sourij, MD, Principal Investigator — Medical University of Graz, Auenbruggerplatz 15
Locations (1):
- Dept. of Internal Medicine, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tripolt NJ, Aberer F, Url J, Hogenauer C, Schreiber F, Eherer A, Sourij C, Obermayer AM, Stadlbauer V, Svehlikova E, Brunner M, Kojzar H, Pferschy PN, Pieber TR, Sourij H. Impact of Duodeno-Jejunal Bypass Liner (EndoBarrierTM) Implantation on Insulin Sensitivity in Patients with Type 2 Diabetes Mellitus (T2DM): A Study Protocol for a Pilot Trial. Diabetes Ther. 2019 Feb;10(1):299-309. doi: 10.1007/s13300-018-0540-z. Epub 2018 Dec 11. PMID 30539524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the University Hospital Graz (LKH-Univ. Klinikum Graz) between January 2016 and September 2016. The first participant was enrolled in February 2016 and the last participant was enrolled in October 2016.
Pre-assignment Details: 11 participants were screened. Due to 1 withdrawal of informed consent 10 participants were enrolled in the trial and got the endobarrier device implanted.
Period: Overall Study
Arm/Group | EndoBarrier
Started | 10 (10 participants started the active study phase)
Implantation of the Endobarrier Device | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EndoBarrier
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 10
Body weight [Mean (Standard Deviation); unit: kilogram] | 121.2 (18.5)
Height [Mean (Standard Deviation); unit: meter] | 1.68 (0.1)
BMI [Mean (Standard Deviation); unit: kilograms divided by height in meters sq] | 43.3 (5.0)
Waist circumference [Mean (Standard Deviation); unit: centimeter] | 128 (12)
Hip circumference [Mean (Standard Deviation); unit: centimeter] | 128 (9)
Waist to hip ratio [Mean (Standard Deviation); unit: Ratio] | 1 (0.1)
systolic blood pressure [Mean (Standard Deviation); unit: millimeters of mercury] | 133 (19)
diastolic blood pressure [Mean (Standard Deviation); unit: millimeters of mercury] | 88 (12)
Diabetes duration in years [Mean (Standard Deviation); unit: years] | 7 (6)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Insulin Sensitivity
Description: insulin sensitivity: measured by mean glucose infusion rate (in a hyperinsulinaemic-euglycaemic clamp) (value at 9 months minus value at baseline)
Time Frame: Baseline and 9 months
Measure: Mean (Standard Deviation); unit: milligram per kilogram per minute
Arm/Group | EndoBarrier
Number analyzed (Participants) | 10
milligram per kilogram per minute | 0.97 (1.36)
Statistical Analysis 1: Comparison: EndoBarrier; The threshold for statistical significance was p = 0.05; Test type: Superiority; p = 0.001, Mixed Models Analysis

2. Secondary Outcome: Changes in Glucagon Like Peptide -1 Levels
Description: Glucagon like peptide -1 levels measured before the Meal Tolerance Test (value at 9 months minus value at baseline)
Time Frame: Baseline and 9 months
Measure: Mean (Standard Deviation); unit: picomole per Liter
Arm/Group | EndoBarrier
Number analyzed (Participants) | 10
picomole per Liter | 18.2 (11.4)
Statistical Analysis 1: Comparison: EndoBarrier; Test type: Superiority; p = 0.081, Friedman test — The threshold for statistical significance was p = 0.05

3. Secondary Outcome: Changes in Gut Permeability
Description: Gut permeability measured by the Lactulose/Mannitol Test (value at 9 months minus value at baseline)
Time Frame: Baseline and 9 months
Measure: Mean (Standard Deviation); unit: lactulose to mannitol ratio
Arm/Group | EndoBarrier
Number analyzed (Participants) | 10
lactulose to mannitol ratio | 0.0039 (0.072)
Statistical Analysis 1: Comparison: EndoBarrier; Test type: Superiority; p = 0.114, Friedman test — The threshold for statistical significance was p = 0.05

4. Secondary Outcome: Changes in Weight
Description: Dual-energy X-ray absorptiometry fat mass (value at 9 months minus value at baseline)
Time Frame: Baseline and 9 months
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | EndoBarrier
Number analyzed (Participants) | 10
kilogram | 53.6 (15.2)
Statistical Analysis 1: Comparison: EndoBarrier; Test type: Superiority; p = 0.021, Friedman test — The threshold for statistical significance was p = 0.05

5. Secondary Outcome: Changes in UKPDS Risk Score for Coronary Heart Disease
Description: The UKPDS Risk Engine provides risk estimates and 95% confidence intervals, in individuals with type 2 diabetes not known to have heart disease, for non-fatal coronary heart disease These can be calculated for any given duration of type 2 diabetes based on current age, sex, ethnicity, smoking status, presence or absence of atrial fibrillation and levels of HbA1c, systolic blood pressure, total cholesterol and HDL cholesterol.
  Units on a scale: 10 year risk to suffer non-fatal coronary heart disease (in %) lower scores mean a better outcome (value at 9 months minus value at baseline)
Time Frame: Baseline and 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EndoBarrier
Number analyzed (Participants) | 10
units on a scale | 16.3 (20.4)
Statistical Analysis 1: Comparison: EndoBarrier; Test type: Superiority; p = 1.00, Friedman test — The threshold for statistical significance was p = 0.05

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | EndoBarrier
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier (N=10)
Dehydration (General disorders) | 1 (1)
duodenal ulcer (Gastrointestinal disorders) | 1 (1)
nausea and vomiting (Gastrointestinal disorders) | 1 (1)
haemorrhoid bleeding (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier (N=10)
Feeling bloated after gastroscopy (Gastrointestinal disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT02769728/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT02769728/SAP_001.pdf